CLINICAL TRIAL: NCT06105814
Title: Improved Diagnostics, Treatment and Follow-up of Acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPEXNOR)
Brief Title: Improved Diagnostics, Treatment and Follow-up of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: COPEXNOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DS-INF-COPEXNOR
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation; Pneumonia; Respiratory Tract Infections
MeSH Terms: conditions — Pneumonia; Respiratory Tract Infections | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Intervention Model Description: COPEXNOR is a prospective, randomized controlled trial with two arms: (1) Standard microbiological diagnostics, with nasopharyngeal swab and induced sputum or endotracheal aspirate for real-time polymerase chain reaction (PCR) and culture, blood cultures and urinary antigen tests, and (2) in addition to (i), induced sputum or endotracheal aspirate analyzed with multiplex PCR (FilmArray).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diagnostics (No Intervention): Standard microbiological diagnostics, with nasopharyngeal swab and induced sputum or endotracheal aspirate for real-time polymerase chain reaction (PCR) and culture, blood cultures and urinary antigen tests
- Rapid diagnostics (Experimental): In addition to standard diagnostics, induced sputum or endotracheal aspirate analyzed with multiplex PCR (FilmArray).
  Interventions: Device: Rapid diagnostics

INTERVENTIONS:
Device: Rapid diagnostics — Sputum sampes will in addition to standard diagnostics be investigated using a rapid diagnostic plattform (FilmArray)
  Arms: Rapid diagnostics

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic and often progressive pulmonary disease, where inflammation and recurrent infections are key pathophysiological contibutors in disease progression. Acute exacerbations of COPD (AECOPD) are often treated with antibiotics, even though only about 50% are caused by bacteria, and the evidence for benefit of empiric antibiotic treatment in AECOPD is conflicting. Microbiological sampling is often insufficient in the setting of AECOPD, and there is a lack of biomarkers distinguishing AECOPD caused by bacteria from those not caused by bacteria, leaving the clinician with few tools to guide the use of antibiotics. Overuse of antibiotics is the main driver of antimicrobial resistance (AMR), a major global public health threat, and obtaining the correct microbiological diagnose is important in guiding treatment of AECOPD.

COPEXNOR seeks to examine which samples give the highest microbiological yield in AECOPD, comparing induced sputum to nasopharyngeal swabs. We will also compare conventional microbiological diagnostics to modern rapid molecular microbiological tests, to evaluate if faster microbiological diagnosis improves antibiotic stewardship. The study aims to define the microbiological etiology causing AECOPD in the Norwegian COPD-population, and examine the lung microbiome over time. COPEXNOR will explore biomarkers in sputum and blood that can be useful for differentiating patients who will benefit from antibiotic treatment from patients who will not.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to the emergency room with a tentative diagnosis of AECOPD, and at least two of the following criteria, more than the daily variation,

  * Increased dyspnea
  * Increased cough
  * Increased sputum production
  * Need for change in medication due to AECOPD
* Signed informed consent. Among patients with temporal or permanent reduced ability to consent, close relatives and/or family members must be asked and may approve or reject participation on behalf of the patient. In cases where close relatives/family members are not available, study personnel may include patients according to conscious judgment.
* Patients will be informed about the study and included by dedicated and approved study personnel (study nurses or study doctors), not by the treating health personnel.

Exclusion Criteria:

* Pulmonary embolism, segmental or larger
* Refractory septic shock (meeting the Sepsis-3 definition of septic shock, and requiring vasopressors ≥ 0.5 mcg/kg/min noradrenaline or equivalent dose of other vasopressor(s)
* Glasgow Coma Scale score 3
* Patients not eligible for lower airways sampling within the first 24 hours of admission
* Palliative situation with life expectancy < 1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Improve microbiological sampling strategies in AECOPD. | Within months to a year after study completion.
  Proportion of AECOPD with a microbiologically verified diagnosis from sputum versus nasopharyngeal swab.
Improve microbiological diagnostic workflow for faster initiation of adequate antibiotic therapy. | Within months to a year after study completion.
  Time to targeted antimicrobial therapy in hours.
Reduce the use of unnecessary broad antimicrobial therapy. | Within months to a year after study completion.
  Proportion of patients with AECOPD who receive targeted antimicrobial therapy.
Increase knowledge of the microbiological etiology in AECOPD. | Within months to a year after study completion.
  Microbiological etiology in AECOPD.
Increased understanding of the lung microbiome over time. | 2-5 years after study completion
  Identify differences in lung microbiome over time, both in AECOPD and stabile state.
Biomarkers at protein level | 2-5 years after study completion
  Identifying biomarkers in blood and sputum that can help differentiate between bacterial and non-bacterial AECOPD
Protein markers of the iron metabolism | 2-5 years after study completion
  Identifying dynamics in iron metabolism in light of etiology.
Biomarkers at the transcriptional level | 2-5 years after study completion
  Identifying different transcriptomic profiles in different causes of AECOPD
Biomarkers for predicting outcome | 2-5 years after study completion
  Identifying biomarkers that can predict outcome in AECOPD.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Heggelund, MD, PhD, Principal Investigator — Medical department, Drammen hospital, Vestre Viken. Department of clinical science, faculty of medicine, University of Bergen.; Karl Erik Müller, MD, PhD, Study Director — Medical department, Drammen hospital, Vestre Viken. Department of clinical science, faculty of medicine, University of Bergen.

IPD SHARING:
Plan to Share IPD: No
Research data is likely to be made avaliable upon reasonable request. It has to be anonymized due to national regulations.